CLINICAL TRIAL: NCT01707849
Title: An Unicenter, Prospective, Randomized, Pilot Study Comparing the Effect of Everolimus-containing Versus mTOR Inhibitor Free Immunosuppression in the Evolution of Hepatitis C Fibrosis After Liver Transplantation.
Brief Title: The Impact of Everolimus Based Immunosuppression in the Evolution of Hepatitis C Fibrosis After Liver Transplantation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Cristina Dopazo Taboada, Liver Surgery and Transplants Consultant, PhD/MD, Hospital Vall d'Hebron
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EVL-VHC-HVH.12
Record Dates: First submitted 2012-10-13; First posted 2012-10-16 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2016-08

CONDITIONS: Hepatitis C Recurrence After Liver Transplant
Keywords: Hepatitis C; Liver Fibrosis; m-TOR inhibitors
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis | interventions — Everolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MMF arm (Active Comparator): MMF arm (n=20)
  They will receive immunosuppression as stipulated by hospital protocol:
  Tacrolimus (levels 8-10ng/mL) and Mycophenalate mofetil 1mg bid(levels 1-3ng/mL).
  Interventions: Drug: MMF arm
- EVL arm (Experimental): EVL arm (n=20):
  Tacrolimus (levels 8-10ng/ml) + everolimus 1mg bid (levels 2-4 ng/mL)
  Interventions: Drug: EVL arm

INTERVENTIONS:
Drug: EVL arm — Patients will be randomized at day 28th post-transplant. This group will receive Tacrolimus+Everolimus.
  Other Names: Everolimus
  Arms: EVL arm
Drug: MMF arm — Patients will be randomized at day 28th post-transplant. This group will continue of current immunosuppressive regimen (Tacrolimus+MMF) / no everolimus introduction.
  Other Names: Mofetil Mycophenolate
  Arms: MMF arm

SUMMARY:
Background:

Hepatitis C recurrence, which invariably occurs in viremic liver transplant (LT) recipients, associated with accelerated liver fibrosis leading to established graft cirrhosis in 40-20% of patients in 5 years with another 5% experiencing an aggressive form with cirrhosis and graft loss in 1 year. Since treatment after LT has a low efficacy, the overall survival of HCV-infected LT recipients is shorter than that of uninfected LT patients.

New immunosuppressive agents such as mTOR inhibitors (Everolimus/Sirolimus) reduce the risk of liver graft rejection, have antifibrotic properties and do not worsen HCV recurrence. Moreover new directly-acting antiviral agents have increased efficacy of interferon-based treatment but their use in LT recipients may be limited by side effects.

Hypothesis:

Use of individualized immunosuppressive regimen and early personalized anti-viral treatment based on recipient and viral factors would improve outcome of HCV infected liver transplant recipients.

Objectives:

1. To evaluate safety and efficacy of two steroid-free immunosuppressive regimens to reduce hepatitis C recurrence associated to fibrosis progression (F≥2 under ISHAK score) at one year post-transplant.
2. To identify viral and recipient factors associated with liver fibrosis progression using ultra-deep pyrosequencing (UDPS).

DETAILED DESCRIPTION:
Study design:

A pilot, open-label, prospective, randomized and unicenter study. As pilot study, the number of patients expected to be included is n=40.

Inclusion criteria:

* Age≥18 years
* First liver transplant
* RNA-HCV positive within 12 months previous to the transplant

Exclusion criteria:

* Multiorgan transplant
* Split liver
* ABO incompatible
* HIV positive patients
* Glomerular Filtration rate ≤60mL/min/1.73m2

Patients will receive double immunosuppression therapy at induction with tacrolimus (basal dose 0.1 mg/Kg/day) and mycophenolate mofetil (MMF, basal dose 2g/day) within the first 12 hours after skin closure.

Patients will be randomized in one of the following groups at day 28th post-transplant:

1. MMF group (n=20): tacrolimus (levels 8-10ng/ml) and MMF (levels 1-3ng/mL).
2. EVL group (n=20): tacrolimus (levels 8-10ng/ml) and everolimus (levels 2- 4 ng/mL).

HCV monitorization:

* HVC-RNA detection and quantification. Serum samples will be taken immediately before liver transplantation, in the anhepatic phase, at the beginning and at the end of the reperfusion, and at 1h, 4h, 8h, 12h, 18h, 1d, 3d, 7d, 14d, 28d, 2m, 3m, 6m, 9m and 12m. Blood samples will be taken from the peripheral circulation and centrifugated within 2 to 3 hours after extraction, aliquoted, and frozen at -80 ºC. The concentration of HCV-RNA will be determined by using a quantitative reverse-transcription polymerase chain reaction (RT-PCR) assay (Cobas Ampliprep/Cobas TaqMan; Roche Molecular Diagnostics, Barcelona, Spain) that achieves a sensitivity of 15 UI/mL and ultra deep pyrosequencing (UDSP) protocols will be used to study DNA genomic factor and viral RNA variability.
* Serum fibrosis markers. Serum samples will be taken at 3rd, 6th and 12th months post-transplant from peripheral circulation and frozen at -21ºC. Serum markers (HA, PIIINP, and TIMP-1) will be analyzed by a fully automated, two-site sandwich immunoassay using direct chemiluminometric technology (ADVIA Centayr XP, Siemens Healthcare Diagnositics). The algorithm including the three markers (3-M-ALG) {score= -7,412 + [ln (HA)x0,681] + [ln (PIIINP)x0.775] + [ln (TIMP-1)]x0,494} will be also obtained.
* Transient elastography (FibroScan). Liver stiffness measurements using Fibroscan (Echosens, Paris, France) will be performed in clinics at 6th and 12th months post-transplant.
* Liver biopsy. Liver biopsy will be performed at 12th months post-transplant. All biopsy specimens will be read by a single pathologist. Necroinflammatory activity and fibrosis stage will be scored using ISHAK classification.

Follow-up and clinical data:

After discharge, patients will be visited in the outpatient clinic monthly for the first 3 months and every 3 months thereafter during the first 12 months post-transplant, at which time clinical and analytical variables will be recorded.Baseline characteristics, HCV genotype and viral load before transplant, surgical variables (type of liver transplant, donor age and steatosis, ischemia time), post-transplantation information and follow-up will be prospectively collected in an electronic database.

Patient withdrawal:

* No consent form given by the patient
* Severe adverse events related to immunosuppressors used
* Steroids are required for long period of time
* Antiviral therapy given before during the first year post-transplant
* Lost follow-up
* Patient death

ELIGIBILITY:
Inclusion Criteria:

* Age≥18 years
* First liver transplant
* RNA-HCV positive within 12 months previous to the transplant

Exclusion Criteria:

* Multiorgan transplant
* Split liver
* Fulminant hepatitis
* ABO incompatible
* HIV positive patients
* Glomerular Filtration rate ≤60mL/min/1.73m2

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
To compare the liver fibrosis progression (F≥2 under ISHAK score) in patients who receive everolimus vs mTOR free immunosuppression | One year
  Liver biopsy will be performed at 12th months post-transplant. All biopsy specimens will be read by a single pathologist. Necroinflammatory activity and fibrosis stage were scored using ISHAK classification.

SECONDARY OUTCOMES:
To identify viral and recipient molecular predictors of fibrosis and anti-HCV treatment responses in liver transplant recipients under steroid-free immunosuppression | Immediately before liver transplantation, in the anhepatic phase, at the beginning and at the end of the reperfusion, and at 1h, 4h, 8h, 12h, 18h, 1dy, 3dy, 7dy, 14dy, 28dy, 2mo, 3mo, 6mo, 9mo and 12mo post-transplant
  Serum samples from the recipient will be taken immediately before liver transplantation, in the anhepatic phase, at the beginning and at the end of the reperfusion, and at 1h, 4h, 8h, 12h, 18h, 1d, 3d, 7d, 14d, 28d, 2m, 3m, 6m, 9m and 12m. Blood samples will be taken from the peripheral circulation and centrifugated within 2 to 3 hours after extraction, aliquoted, and frozen at -80 ºC.
  * The concentration of HCV-RNA will be determined by using a quantitative reverse-transcription polymerase chain reaction (RT-PCR) assay (Cobas Ampliprep/Cobas TaqMan; Roche Molecular Diagnostics, Barcelona, Spain) that achieves a sensitivity of 15 UI/mL. -
  * DNA will be extracted from the liver donor and the recipient to characterize DNA polymorphisms. RNA Viral population complexity and presence of resistant mutations will be also studied using ultra-deep pyrosequence using eithre GS-Junior or GS-FLX platforms

OTHER OUTCOMES:
To analyze liver fibrosis progression using serum markers | 3rd, 6th and 12th months post-transplant
  Serum samples will be taken from peripheral circulation an frozen at -21ºC. Serum markers (HA, PIIINP, and TIMP-1) are analyzed by a fully automated, two-site sandwich immunoassay using direct chemiluminometric technology (ADVIA Centayr XP, Siemens Healthcare Diagnositics). The algorithm including the three markers (3-M-ALG) {score= -7,412 + [ln (HA)x0,681] + [ln (PIIINP)x0.775] + [ln (TIMP-1)]x0,494} will be also obtained.
To analyze liver fibrosis progression using liver stiffness | 6th and 12th months post-transplant
  Transient elastography (FibroScan) for liver stiffness measurements will be performed in clinics.
To analyze the incidence of acute rejection and steroid-resistant acute rejection | 6th and 12th months post-transplant
  Rejection will be suspected in patients with an increase in the levels of bilirrubin, transaminases or alkaline phosphatase. Doppler ultrasound will be performed in order to discard biliary dilation and to confirm portal and arterial flow patency. A liver biopsy will be performed and graft rejection will be defined and stratified according to the BANFF criteria.
To analyze the timing to the first acute rejection episode in both study groups | 6th and 12 months post-transplant
To analyze need of antiviral therapy at the end of the first year post-transplant | One year post-transplant
  Antiviral treatment will be considered at the end of the 12-months study period if moderated fibrosis (F≥2 under ISHAK score)is diagnosed and the patient do not have any contraindications to therapy
To analyze graft and patient survival | One year post-transplant
To analyze the incidence of patient withdrawal | One year post-transplant
To analyze the incidence of cardiovascular risk factors | 6th and 12th months post-transplant
  Cardiovascular risk factors will be defined as follow:
  Arterial hypertension. Defined as blood pressure >140/90 mmHg at two following visits according to the European Society of Hypertension criteria.
  Diabetes Mellitus. Defined as fasting plasma glucose > 126 mg/dL at two following visits according to the World Health Organization.
  Dyslipidemia. Defined as hypercholesterolemia > 220mg/dL and hypertriglyceridemia >200mg/dL at two following visits.

CONTACTS AND LOCATIONS:
Overall Officials: Itxarone Bilbao, PhD/MD, Principal Investigator — Department of HPB Surgery and Transplant, Hospital Vall d´Hebron (Barcelona, Spain); Ramon Charco, PhD/MD, Study Director — Department of HPB and Transplants, Hospital Vall d´Hebron (Barcelona, Spain); Josep Quer, PhD/MD, Study Chair — Hepatology Unit, Department of Internal Medicine, Hospital Vall d´Hebron, CIBERehd, Barcelona (Spain); Francisco Rodríguez, PhD/MD, Study Chair — Biochemistry Laboratory, Hospital Vall d´Hebron, Barcelona (Spain); Gonzalo Sapisochin, PhD/MD, Study Chair — Department of HPB Surgery and Transplant, Hospital Vall d´Hebron, Barcelona (Spain); Lluis Castells, PhD/MD, Study Chair — Hepatology Unit, Department of Internal Medicine, Hospital Vall d´Hebron, CIBERehd, Barcelona (Spain); Isabel Campos, PhD, Study Chair — Hepatology Unit, Department of Internal Medicine, Hospital Vall d´Hebron, CIBERehd, Barcelona (Spain); Helena Allende, PhD/MD, Study Chair — Department of Anatomo-Pathology, Hospital Vall d´Hebron, Barcelona (Spain); Jose Luis Lazaro, PhD, Study Chair — Department of HPB surgery and Transplant, Hospital Vall d´Hebron, Barcelona (Spain); Cristina Dopazo-Taboada, PhD/MD, Study Chair — Department of HPB and Transplant, Hospital Vall d´Hebron, Barcelona (Spain)
Locations (1):
- Department of HPB Surgery and Transplant, Hospital Vall d´Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biecker E, De Gottardi A, Neef M, Unternahrer M, Schneider V, Ledermann M, Sagesser H, Shaw S, Reichen J. Long-term treatment of bile duct-ligated rats with rapamycin (sirolimus) significantly attenuates liver fibrosis: analysis of the underlying mechanisms. J Pharmacol Exp Ther. 2005 Jun;313(3):952-61. doi: 10.1124/jpet.104.079616. Epub 2005 Mar 15. PMID 15769867
- [Background] Neef M, Ledermann M, Saegesser H, Schneider V, Reichen J. Low-dose oral rapamycin treatment reduces fibrogenesis, improves liver function, and prolongs survival in rats with established liver cirrhosis. J Hepatol. 2006 Dec;45(6):786-96. doi: 10.1016/j.jhep.2006.07.030. Epub 2006 Sep 22. PMID 17050028
- [Background] Patsenker E, Schneider V, Ledermann M, Saegesser H, Dorn C, Hellerbrand C, Stickel F. Potent antifibrotic activity of mTOR inhibitors sirolimus and everolimus but not of cyclosporine A and tacrolimus in experimental liver fibrosis. J Hepatol. 2011 Aug;55(2):388-98. doi: 10.1016/j.jhep.2010.10.044. Epub 2010 Dec 17. PMID 21168455
- [Background] Bilbao I, Sapisochin G, Dopazo C, Lazaro JL, Pou L, Castells L, Caralt M, Blanco L, Gantxegi A, Margarit C, Charco R. Indications and management of everolimus after liver transplantation. Transplant Proc. 2009 Jul-Aug;41(6):2172-6. doi: 10.1016/j.transproceed.2009.06.087. PMID 19715864
- [Background] Wagner D, Kniepeiss D, Schaffellner S, Jakoby E, Mueller H, Fahrleitner-Pammer A, Stiegler P, Tscheliessnigg KH, Iberer F. Sirolimus has a potential to influent viral recurrence in HCV positive liver transplant candidates. Int Immunopharmacol. 2010 Aug;10(8):990-3. doi: 10.1016/j.intimp.2010.05.006. Epub 2010 May 17. PMID 20483386
- [Background] McKenna GJ, Trotter JF, Klintmalm E, Onaca N, Ruiz R, Jennings LW, Neri M, O'Leary JG, Davis GL, Levy MF, Goldstein RM, Klintmalm GB. Limiting hepatitis C virus progression in liver transplant recipients using sirolimus-based immunosuppression. Am J Transplant. 2011 Nov;11(11):2379-87. doi: 10.1111/j.1600-6143.2011.03767.x. Epub 2011 Oct 3. PMID 21967703
- [Background] Carrion JA, Torres F, Crespo G, Miquel R, Garcia-Valdecasas JC, Navasa M, Forns X. Liver stiffness identifies two different patterns of fibrosis progression in patients with hepatitis C virus recurrence after liver transplantation. Hepatology. 2010 Jan;51(1):23-34. doi: 10.1002/hep.23240. PMID 19839063
- [Background] Pungpapong S, Nunes DP, Krishna M, Nakhleh R, Chambers K, Ghabril M, Dickson RC, Hughes CB, Steers J, Nguyen JH, Keaveny AP. Serum fibrosis markers can predict rapid fibrosis progression after liver transplantation for hepatitis C. Liver Transpl. 2008 Sep;14(9):1294-302. doi: 10.1002/lt.21508. PMID 18756457
- [Background] Nobili V, Parkes J, Bottazzo G, Marcellini M, Cross R, Newman D, Vizzutti F, Pinzani M, Rosenberg WM. Performance of ELF serum markers in predicting fibrosis stage in pediatric non-alcoholic fatty liver disease. Gastroenterology. 2009 Jan;136(1):160-7. doi: 10.1053/j.gastro.2008.09.013. Epub 2008 Sep 20. PMID 18992746
- [Background] Carrion JA, Fernandez-Varo G, Bruguera M, Garcia-Pagan JC, Garcia-Valdecasas JC, Perez-Del-Pulgar S, Forns X, Jimenez W, Navasa M. Serum fibrosis markers identify patients with mild and progressive hepatitis C recurrence after liver transplantation. Gastroenterology. 2010 Jan;138(1):147-58.e1. doi: 10.1053/j.gastro.2009.09.047. Epub 2009 Sep 26. PMID 19786026
- [Background] Garcia-Retortillo M, Forns X, Feliu A, Moitinho E, Costa J, Navasa M, Rimola A, Rodes J. Hepatitis C virus kinetics during and immediately after liver transplantation. Hepatology. 2002 Mar;35(3):680-7. doi: 10.1053/jhep.2002.31773. PMID 11870384
- [Background] Domingo E, Gomez J. Quasispecies and its impact on viral hepatitis. Virus Res. 2007 Aug;127(2):131-50. doi: 10.1016/j.virusres.2007.02.001. Epub 2007 Mar 8. PMID 17349710
- [Background] Martell M, Esteban JI, Quer J, Genesca J, Weiner A, Esteban R, Guardia J, Gomez J. Hepatitis C virus (HCV) circulates as a population of different but closely related genomes: quasispecies nature of HCV genome distribution. J Virol. 1992 May;66(5):3225-9. doi: 10.1128/JVI.66.5.3225-3229.1992. PMID 1313927
- [Background] Vignuzzi M, Stone JK, Arnold JJ, Cameron CE, Andino R. Quasispecies diversity determines pathogenesis through cooperative interactions in a viral population. Nature. 2006 Jan 19;439(7074):344-8. doi: 10.1038/nature04388. Epub 2005 Dec 4. PMID 16327776
- [Background] Forns X, Purcell RH, Bukh J. Quasispecies in viral persistence and pathogenesis of hepatitis C virus. Trends Microbiol. 1999 Oct;7(10):402-10. doi: 10.1016/s0966-842x(99)01590-5. PMID 10498948
- [Background] Wang GP, Sherrill-Mix SA, Chang KM, Quince C, Bushman FD. Hepatitis C virus transmission bottlenecks analyzed by deep sequencing. J Virol. 2010 Jun;84(12):6218-28. doi: 10.1128/JVI.02271-09. Epub 2010 Apr 7. PMID 20375170
- [Background] Bull RA, Luciani F, McElroy K, Gaudieri S, Pham ST, Chopra A, Cameron B, Maher L, Dore GJ, White PA, Lloyd AR. Sequential bottlenecks drive viral evolution in early acute hepatitis C virus infection. PLoS Pathog. 2011 Sep;7(9):e1002243. doi: 10.1371/journal.ppat.1002243. Epub 2011 Sep 1. PMID 21912520
- [Background] Thomas DL, Thio CL, Martin MP, Qi Y, Ge D, O'Huigin C, Kidd J, Kidd K, Khakoo SI, Alexander G, Goedert JJ, Kirk GD, Donfield SM, Rosen HR, Tobler LH, Busch MP, McHutchison JG, Goldstein DB, Carrington M. Genetic variation in IL28B and spontaneous clearance of hepatitis C virus. Nature. 2009 Oct 8;461(7265):798-801. doi: 10.1038/nature08463. PMID 19759533
- [Background] Afdhal NH, McHutchison JG, Zeuzem S, Mangia A, Pawlotsky JM, Murray JS, Shianna KV, Tanaka Y, Thomas DL, Booth DR, Goldstein DB; Pharmacogenetics and Hepatitis C Meeting Participants. Hepatitis C pharmacogenetics: state of the art in 2010. Hepatology. 2011 Jan;53(1):336-45. doi: 10.1002/hep.24052. PMID 21254181
- [Background] Ge D, Fellay J, Thompson AJ, Simon JS, Shianna KV, Urban TJ, Heinzen EL, Qiu P, Bertelsen AH, Muir AJ, Sulkowski M, McHutchison JG, Goldstein DB. Genetic variation in IL28B predicts hepatitis C treatment-induced viral clearance. Nature. 2009 Sep 17;461(7262):399-401. doi: 10.1038/nature08309. Epub 2009 Aug 16. PMID 19684573
- [Background] Suppiah V, Moldovan M, Ahlenstiel G, Berg T, Weltman M, Abate ML, Bassendine M, Spengler U, Dore GJ, Powell E, Riordan S, Sheridan D, Smedile A, Fragomeli V, Muller T, Bahlo M, Stewart GJ, Booth DR, George J. IL28B is associated with response to chronic hepatitis C interferon-alpha and ribavirin therapy. Nat Genet. 2009 Oct;41(10):1100-4. doi: 10.1038/ng.447. Epub 2009 Sep 13. PMID 19749758
- [Background] Tanaka Y, Nishida N, Sugiyama M, Kurosaki M, Matsuura K, Sakamoto N, Nakagawa M, Korenaga M, Hino K, Hige S, Ito Y, Mita E, Tanaka E, Mochida S, Murawaki Y, Honda M, Sakai A, Hiasa Y, Nishiguchi S, Koike A, Sakaida I, Imamura M, Ito K, Yano K, Masaki N, Sugauchi F, Izumi N, Tokunaga K, Mizokami M. Genome-wide association of IL28B with response to pegylated interferon-alpha and ribavirin therapy for chronic hepatitis C. Nat Genet. 2009 Oct;41(10):1105-9. doi: 10.1038/ng.449. Epub 2009 Sep 13. PMID 19749757
- [Background] Smith KR, Suppiah V, O'Connor K, Berg T, Weltman M, Abate ML, Spengler U, Bassendine M, Matthews G, Irving WL, Powell E, Riordan S, Ahlenstiel G, Stewart GJ, Bahlo M, George J, Booth DR; International Hepatitis C Genetics Consortium (IHCGC). Identification of improved IL28B SNPs and haplotypes for prediction of drug response in treatment of hepatitis C using massively parallel sequencing in a cross-sectional European cohort. Genome Med. 2011 Aug 31;3(8):57. doi: 10.1186/gm273. PMID 21884576